CLINICAL TRIAL: NCT00731146
Title: Effects of Ultrasound Guidance on the Minimum Effective Anesthetic Volume Required for Interscalene Brachial Plexus Block Versus Nerve Stimulator Guidance
Brief Title: Effects of Technique on the Local Anesthetic Dose Required for Interscalene Brachial Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Dr. Colin McCartney, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHSCA02
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Arthroscopic Shoulder Surgery
Keywords: Interscalene Brachial Plexus Block; Regional Anesthesia; Ultrasound guided peripheral nerve block; Minimum Effective Anesthetic Volume; Nerve Stimulator guided peripheral nerve block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Ultrasound (Active Comparator): Participants will receive an ultrasound guided interscalene brachial plexus block
  Interventions: Other: Ultrasound Minimum Effective Anesthetic Volume
- 2 - Nerve Stimulator (Active Comparator): Participants will receive a nerve stimulator guided interscalene brachial plexus block
  Interventions: Other: Nerve Stimulator Minimum Effective Anesthetic Volume

INTERVENTIONS:
Other: Ultrasound Minimum Effective Anesthetic Volume — Each sequential participant in this group will be assigned a dose based on the success or failure of the previous participant's block. The starting dose will be 10mL of 0.5% ropivacaine. Each success will decrease the dose by 2.5mL and each failure will subsequently increase the dose by 2.5mL.
  Arms: 1 - Ultrasound
Other: Nerve Stimulator Minimum Effective Anesthetic Volume — Each sequential participant in this group will be assigned a dose based on the success or failure of the previous participant's block. The starting dose will be 10mL of 0.5% ropivacaine. Each success will decrease the dose by 2.5mL and each failure will subsequently increase the dose by 2.5mL.
  Arms: 2 - Nerve Stimulator

SUMMARY:
Interscalene brachial plexus block (ISBPB) is a common nerve block given to patients who are undergoing shoulder surgery. This block has a low, but still significant, rate of complications. Reducing the volume of local anesthetic given during the block may allow some of these complications to be avoided. Participants will be randomly assigned to a group to undergo ISBPB under ultrasound or nerve stimulator guidance. Each group will initially receive 10mL of local anesthetic. The volume used for each subsequent patient depends upon the success or failure of the previous patient's block - a failure will cause the volume given to increase by 2.5mL, while a success will cause the volume to decrease by the same amount. We hypothesize that the minimum effective anesthetic volume in 50% of patients will be significantly lower in the ultrasound guided group than in the nerve stimulator group. We further hypothesize that this lower volume will lead to a decreased rate of complications.

DETAILED DESCRIPTION:
This will be a randomized, single-blind, up-down sequential allocation study. Patients will be randomly assigned to one of two groups, and receive either an ultrasound-guided or nerve-stimulator guided interscalene brachial plexus block. The initial local anesthetic volume in both groups will be 10mL. The outcome of each patient's block will determine the dose for the subsequent patient. When an effective ISBPB is observed, as defined by a NRS (patient-rated pain on a scale from 0 to 10) rating of 0 within 30 minutes post-surgery, the volume of local anesthetic solution used for the next patient will be decreased by 2.5mL. Conversely, when an ineffective ISBPB is observed, the volume of local anesthetic used for the next patient will be increased by 2.5mL.

The goal of this study is to determine the minimum effective anesthetic volume of ropivacaine 0.5% providing analgesia in patients when using either ultrasound or a nerve stimulator to guide placement of the block. The primary outcome measure will be the pain score of the patient on a numeric rating score during the 30 minutes after surgery.

A number of previous studies have suggested that ultrasound-guidance is beneficial for peripheral nerve blocks in terms of block performance time, success rates, and block quality. Some studies have also shown that ultrasound-guidance can reduce the volume of local anesthetic needed to perform a successful block. This study may reveal that less local anesthetic is needed under ultrasound guidance than under nerve stimulator, which may potentially reduce some of the common complications of ISBPB.

We hypothesize that ISBPB done under ultrasound guidance will have a lower minimum effective local anesthetic volume than ISBPB done under nerve stimulation. Further, we hypothesize that the lower volume will reduce the incidence of some of the complications of ISBPB.

Using lower volumes of local anesthetic while still maintaining effective analgesia may reduce some of the common complications of ISBPB. It may also allow this beneficial analgesic technique to be given to patients with some respiratory risk factors who are currently unable to receive it.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving interscalene brachial plexus block for arthroscopic shoulder surgery

Exclusion Criteria:

* ASA >III, and body mass index (BMI) >35, pre-existing chronic obstructive pulmonary disease (COPD), unstable asthma, psychiatric history, renal or hepatic impairment, allergy to ropivacaine, and opioid tolerance (>30 mg oral morphine or equivalent per day).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-02 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Pain Rating as based on 11 point NRS scale | within 30 minutes or less post-surgery

SECONDARY OUTCOMES:
Diaphragmatic Function (as assessed by diaphragmatic movement on ultrasound) | within 30 minutes post-block

CONTACTS AND LOCATIONS:
Overall Officials: Colin J McCartney, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada